CLINICAL TRIAL: NCT02310373
Title: Effects of Nicotine-Free Hookah Smoking on Blood Flow to the Heart, Muscle and Skin
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Responsible Party/PI passed away. All subjects enrolled completed study prior to termination.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00037529
Record Dates: First submitted 2014-11-25; First posted 2014-12-08 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Nicotine-free Hookah Smoking
Keywords: Nicotine-free hookah; Waterpipe; Smoking; Sympathetic
MeSH Terms: conditions — Water Pipe Smoking; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicotine free hookah (herbal/steam stones) smoking (Experimental): Healthy habitual Hookah smokers will undergo microneurography, myocardial contrast echocardiogram or venous occlusion plethysmography before and after nicotine free hookah smoking.
  Interventions: Other: Nicotine free hookah smoking

INTERVENTIONS:
Other: Nicotine free hookah smoking — Subjects will smoke waterpipe in a controlled research environment

SUMMARY:
This is a pilot study on the acute effects of nicotine-free hookah (herbal/steam stones) smoking on the sympathetic neural control of the human cardiovascular system. Hookah smoking is known to transiently increase blood pressure and heart rate while decreasing heart rate variability suggesting - but not proving - sympathetic mediation. The contribution of nicotine to these effects is unknown. Here the investigators will directly measure the acute effects of nicotine-free Hookah smoking on sympathetic nerve activity with microneurography (intraneural microelectrodes) and quantify associated regional changes in vasomotor tone.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 39 years of age
* Habitual Hookah smoker defined as having smoked Hookah >=12 times in the past 12 months
* Have not smoked cigarettes within the past 12 months

Exclusion Criteria:

* Exhaled carbon monoxide level greater than 10 ppm* as evidence of current or recent cigarette (excluded if smoked cigarette within 12 months) or Hookah smoking (excluded if smoked Hookah within past 72 hours)
* History of cardiopulmonary disease
* Use of any prescription medication with exception of oral contraceptive pills
* History of psychiatric illness
* History of neurologic disease
* BMI ≥ 35
* Evidence of any of the above by physical examination, ECG or echocardiogram
* Smoked cigarette in the past 12 months
* History of illicit drug use
* Pregnant
* Any other condition(s) deemed by the physician investigators that put subjects at risk for participating in the study

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in sympathetic nerve activity | Change from baseline in sympathetic nerve activity at 1 hr
  Multi-unit recordings of sympathetic nerve activity will be obtained with single-use sterile tungsten microelectrodes inserted selectively into muscle or skin nerve fascicles of the peritoneal nerve.

SECONDARY OUTCOMES:
Change in regional myocardial perfusion | Change from baseline in regional myocardial perfusion at 1 hr
  Myocardial contrast echocardiography will be used to measure regional myocardial perfusion (i.e. capillary blood volume) and coronary flow reserve.

OTHER OUTCOMES:
Change in leg blood flow | Change from baseline in leg blood flow at 1 hr
  Lower leg blood flow will be measured with standard venous occlusion plethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States